CLINICAL TRIAL: NCT04283500
Title: Buprenorphine Loading in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Emergency Medicine Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-01700
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Results first posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-03

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine, Naloxone Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BUP treatment arm (Experimental): Subjects will be given BUP 32mg in 2 doses, and observed for at least 90 minutes after the 2nd dose. The whole process will take a total of about 3-4 hours including the consenting process. Subjects will be asked questions and be examined repeatedly. Subjects will have 4 in-person visits and a phone call in addition to review of medical records.
  Interventions: Drug: Buprenorphine Naloxone

INTERVENTIONS:
Drug: Buprenorphine Naloxone — Participants will receive the BUP SL 32mg in divided doses rather than all at once. If after the initial 8mg dose a participant experiences over-sedation or another adverse event that would preclude further dosing, such as an allergic reaction, the subsequent dose will not be administered and the patient will be withdrawn from the study. The participant will be reassessed for other possible etiologies for these symptoms.
  Other Names: Suboxone

SUMMARY:
Buprenorphine (BUP) is FDA-approved for the treatment of opioid withdrawal and opioid use disorder. Few ED providers have received the necessary DEA registration (aka X waiver) required to prescribe BUP, and urgent appointments to continue ongoing BUP treatment may not be readily available, thus leading to medication discontinuity. A loading dose induction strategy with 32mg of BUP may help effectively link ED patients to outpatient treatment while minimizing known barriers to ED uptake. Administering a "loading dose" of BUP to saturate mu-opioid receptors would extend the duration of action and provide additional time to secure ongoing treatment. Further, BUP's ceiling effect on respiratory depression makes it a remarkably safe drug even at high doses. In recent years, ED providers have begun to incorporate this approach into clinical protocols, however, it has not been formally studied in this clinical setting. The investigator's study represents the necessary step of studying this novel approach in the ED setting to define the parameters for clinical protocols and large-scale studies.

DETAILED DESCRIPTION:
A novel induction strategy, in which a loading dose of Buprenorphine (BUP) 32mg is administered, has the potential to mitigate barriers to treatment initiation. ED providers can treat patients with BUP for opioid withdrawal since DEA registration (X-waiver) is not required unless they wish to issue a prescription. Current BUP induction protocols, developed for inpatient and ambulatory care settings as well as for unobserved self- administration via prescription, usually recommend a first day dose of 8mg given in divided doses of 2- 4mg. However, patients discharged with ≤ 8mg SL total dose may experience return of withdrawal symptoms and/or opioid craving within only 4 hours.Treatment with a loading dose of 32mg in the ED may provide the necessary bridge treatment, relieving symptoms of withdrawal until a patient is able to attend a follow up appointment for further treatment.

ELIGIBILITY:
Inclusion Criteria:

* Is able to speak English sufficiently to understand the study procedures and provide written informed consent to participate in the study.
* Meets DSM-5 criteria for moderate to severe OUD
* Has a positive urine screen for opioids and a negative urine screen for methadone
* Must be experiencing opioid withdrawal with a COWS score ≥8
* Is willing and able to participate in the study and follow study procedures
* Is able to provide adequate and reliable locator information for follow-up
* Has reliable access to a phone

Exclusion Criteria:

* Is currently engaged in medication treatment for OUD with methadone, BUP, or naltrexone
* Has a urine toxicology test that is positive for methadone or buprenorphine
* Currently requires prescribed opioids for treatment of an ongoing pain condition
* Has a known allergy to BUP
* Is pregnant as determined by urine hCG testing at the index ED visit
* Is breastfeeding as determined by self-report
* Has medical, psychiatric, or concurrent substance use conditions or severe cognitive impairment which might prelude safe participation
* Is a prisoner or in police custody at the time of the index ED visit
* Has previously enrolled in the current study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-02-25 (Actual); Study Completion 2023-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ryan McCormack, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data. Upon reasonable request. Requests should be directed to Ryan.McCormack@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BUP Treatment Arm
Started | 15
Completed Day 0 | 14
Completed Day 1 | 14
Completed Day 2 | 13
Completed Day 3 | 11
Completed (Day 30) | 6
Not Completed | 9
Not completed — Lost to Follow-up | 8
Not completed — Withdrawn by study team prior to intervention for not meeting post-enrollment inclusion criteria | 1

BASELINE CHARACTERISTICS:
Arm/Group | BUP Treatment Arm
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (4.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 4
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Rapid Induction
Description: This will be measured by the proportion of participants who report Successful Rapid Induction. Participants will receive a loading dose of BUP SL 32mg in the ED without experiencing a clinically significant serious and/or severe adverse event (AE) related to the intervention - specifically, the receipt of a dose of BUP SL greater than 8mg during the Index ED visit. Successful rapid induction is defined only by the outcome of the participant's visit, and not by any following research visits.
Time Frame: Day 0
Measure: Count of Participants; unit: Participants
Arm/Group | BUP Treatment Arm
Number analyzed (Participants) | 14
Participants | 14

2. Secondary Outcome: Opioid Withdrawal at Conclusion of Index Visit as Measured by the Clinical Opiate Withdrawal Scale (COWS)
Description: The Clinical Opiate Withdrawal Scale (COWS) is an 11-item scale designed to be administered by a clinician. The tool can be used in both inpatient and outpatient settings to reproducibly rate common signs and symptoms of withdrawal and monitor these symptoms over time. The summed score can be used to help clinicians determine the stage or severity of withdrawal and assess the level of physical dependence on opioids. The total score ranges from 0 to 48. The interpretation of scores is as follows: 5-12 = mild; 13-24 = moderate; 25-36 = moderately severe; more than 36 = severe withdrawal.
Time Frame: Index ED Visit 1(Day 0)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | BUP Treatment Arm
Number analyzed (Participants) | 14
score on a scale | 1 [1 to 5]

3. Secondary Outcome: Number of Participants With Withdrawal Suppresion at Day 1 (24 Hours)
Description: Participants who had suppression of opioid withdrawal within 24 hours of receipt of buprenorphine at the index visit as measured by having none of the following: 1) having a COWS score of >7 at the Day 1 research visit, 2) having objective signs of opioid withdrawal as assessed by a medical clinician, or 3) participant self-report of opioid use to treat opioid withdrawal.
Time Frame: Day 1 (24 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | BUP Treatment Arm
Number analyzed (Participants) | 14
Participants | 9

4. Secondary Outcome: Number of Participants With Withdrawal Suppresion by Day 2
Description: Participants who had suppression of opioid withdrawal within 48 hours of receipt of buprenorphine at the index visit as measured by having none of the following: 1) having a COWS score of >7 at the Day 1 research visit, 2) having objective signs of opioid withdrawal as assessed by a medical clinician, or 3) participant self-report of opioid use to treat opioid withdrawal.
Time Frame: Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | BUP Treatment Arm
Number analyzed (Participants) | 12
Participants | 6

5. Secondary Outcome: Number of Participants With Withdrawal Suppression on Day 3
Description: Participants who had suppression of opioid withdrawal within 72 hours of receipt of buprenorphine at the index visit as measured by having none of the following: 1) having a COWS score of >7 at the Day 1 research visit, 2) having objective signs of opioid withdrawal as assessed by a medical clinician, or 3) participant self-report of opioid use to treat opioid withdrawal.
Time Frame: Day 3
Measure: Count of Participants; unit: Participants
Arm/Group | BUP Treatment Arm
Number analyzed (Participants) | 12
Participants | 4

ADVERSE EVENTS:
Time Frame: 1 month
Description: systematic - standard questionnaire and medical record review
Arm/Group | BUP Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 1/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BUP Treatment Arm (N=14)
Diarrhea (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT04283500/Prot_SAP_000.pdf